CLINICAL TRIAL: NCT03942003
Title: Investigation of the Analgesic Effects of the Rhomboid Intercostal Block and Pectoral Nerve Block Applied in Breast Surgery
Brief Title: Analgesic Effects of Rhomboid Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rhomboid
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Pain; Anesthesia
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rhomboid (Experimental): When applying the Rhomboid nerve block, the patient is tilted to the side position so that the corresponding breast is at the top. After T7 up to T10 sterile preparation of the C7 spinous projection, the convex probe shows a rhomboid muscle at the level of T5 and block is applied with 0.25% bupivacaine (20 cc), 2% lidocaine (10 cc) and 10 cc SF mixture.
  Interventions: Procedure: rhomboid blocks
- Pectoral (Experimental): The PEC I field block is performed by administering 10 cc of local anesthetic between the pectoralis minor and the major at the 2nd costal position. PEC II field block is performed using linear USG probe visibly in 3rd and 4th ribs while the patient is in supine position. In this block, a total of 20 cc 0.25% bupivacaine (10 cc), 2% lidocaine (5 cc) and 5 cc SF mixture were used to block the area between the pectoralis minor muscle and the serratus muscle
  Interventions: Procedure: PEC blocks
- Control (Sham Comparator): Infiltration analgesia was performed.
  Interventions: Procedure: Control groups

INTERVENTIONS:
Procedure: rhomboid blocks — Rhomboid nerve block was performed
  Arms: Rhomboid
Procedure: PEC blocks — PEC I-II blocks was performed
  Arms: Pectoral
Procedure: Control groups — Infiltration analgesia was performed
  Arms: Control

SUMMARY:
Breast surgery is a common surgical procedure because of the prevalence of breast cancer. Postoperative analgesia management in breast surgery is difficult due to the content of the surgical procedure and the complex innervation of the breast. Multimodal approach is recommended for postoperative analgesia. Therefore, various methods are used. There was no comparison of these two blocks to control group in the literature. In this study, the investigators planned to investigate the postoperative pain, analgesic usage dose and side effects of patients undergoing breast surgery under general anesthesia with a rhomboid area block, pectoral area block.

DETAILED DESCRIPTION:
Regional methods and pharmacological treatments are among these methods. The blocks of serratus, pectoral and rhomboid from the regional blocks are used more safely and with increasing frequency, especially with the introduction of ultrasonography in the clinic. In 2016, the rhomboid intercostal nerve block was identified and presented in the literature as a case report. In the rhomboid block, the analgesia created by the local anesthetic on the anterior thoracic wall was used. For patients who will undergo elective breast surgery, the routine routinely applied in our clinic is a multimodal approach, which involves conducting a peripheral nerve block following general anesthesia induction for postoperative analgesia. All patients before the block are standardized and intravenous vascular access is opened. In our clinic, all peripheral blocks are performed under sterile conditions accompanied by ultrasound and stimulator. When applying the Rhomboid nerve block, the patient is tilted to the side position so that the corresponding breast is at the top. After T7 up to T10 sterile preparation of the C7 spinous projection, the convex probe shows a rhomboid muscle at the level of T5 and block is applied with 0.25% bupivacaine (20 cc), 2% lidocaine (10 cc) and 10 cc SF mixture. The PEC I field block is performed by administering 10 cc of local anesthetic between the pectoralis minor and the major at the 2nd costal position. PEC II field block is performed using linear USG probe visibly in 3rd and 4th ribs while the patient is in supine position. In this block, a total of 20 cc 0.25% bupivacaine (10 cc), 2% lidocaine (5 cc) and 5 cc SF mixture were used to block the area between the pectoralis minor muscle and the serratus muscle. Sensory block is evaluated with cold stimulus (0 = no cold sensation, 1 = cold feeling severely decreased, 2 = cold feeling slightly reduced, 3 = normal cold feeling). Patients undergoing breast surgery routinely undergo general anesthesia with propofol 2-3 mg / kg, fentanyl 1mcq / kg, lidocaine 1 mg / kg and rocuronium 0.6 mg / kg. The postoperative analgesic needs of the patients will be recorded in the patient-controlled analgesia device. Postoperative pain, digital evaluation scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) of all patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* mastectomy
* general anesthesia

Exclusion Criteria:

* Diabetes mellitus
* Chronic analgesic treatment
* cardiovascular disease
* non-cooperative patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesic consumption | at first 24 hour of postoperative period
  Postoperative analgesic needs of patients will be recorded in the patient-controlled analgesia device. Postoperative pain, digital evaluation scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) of all patients will be recorded.

SECONDARY OUTCOMES:
Sleep quality: NRS | at first morning after operation day
  The postoperative first night sleep quality of the patients will be recorded with NRS (0 = not sleeping all night, 10 = very good sleep).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Siences Diskapi Yildirim Beyazit T&R hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No